CLINICAL TRIAL: NCT02082028
Title: Randomized Clinical Trial on the Efficacy of Self-Monitoring Blood Glucose in the Context of a Chronic Care Model for Type 2 Diabetes Patients Treated With Oral Agents Only
Brief Title: Efficacy of a Chronic Care Model Supported by Self Monitoring of Blood Glucose With BGStar Over Usual Care in Improving Glycemic Control in Patients With Type 2 Diabetes Not Treated With Insulin
Acronym: SELF CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGSTA_L_05978
Record Dates: First submitted 2014-03-06; First posted 2014-03-07 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (BGStar) (Experimental): Patients will be educated within the context of the SINERGIA educational program to understand how to manage their own diabetes on the basis of their Self Monitoring of Blood Glucose values obtained with BGStar. Patients will be requested two 6-points profiles monthly.
  Interventions: Device: BGStar
- B (traditional approach) (Active Comparator): Usual approach for the disease management. Patients in Group B will receive usual education and, at any time during the study duration, if needed, will be instructed on Self Monitoring of Blood Glucose, performed with any glucose meter.
  Interventions: Device: glucose meter

INTERVENTIONS:
Device: BGStar
  Arms: A (BGStar)
Device: glucose meter
  Arms: B (traditional approach)

SUMMARY:
To demonstrate the superiority of a chronic care model (SINERGIA model) supported by the Self Monitoring of Blood Glucose with BGStar over usual care in improving glycemic control at 12 months in patients with type 2 diabetes not treated with insulin.

DETAILED DESCRIPTION:
The planned study duration is 36 months (9 quarters). The estimated duration of screening/enrollment will be 12 months, followed by the 12-month experimental phase, plus the 12-month follow-up in the observational phase.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age ≥ 45 years
* Type 2 diabetes
* First access at the diabetes clinic
* Any diabetes duration
* HbA1c >7.0 and ≤ 9.0%
* Already treated with any oral antidiabetic agent (OAD) or requiring the initiation of therapy with OAD
* Patients not using SMBG or using SMBG with a frequency ≤1 test/week
* Written informed consent

Exclusion Criteria:

Treatment with insulin or need to start insulin regimens or continuous sub-cutaneous insulin infusion at the first access; Refusal or inability to give informed consent to participate in the study;

Conditions / situations such as:

* Patients with short life expectancy;
* Patients with conditions/concomitant diseases making them non evaluable for the primary efficacy endpoint according to physician's judgment;
* Requirement for concomitant treatment that could bias primary evaluation (i.e. corticosteroid treatment);
* Patient is the Investigator or any Sub-Investigator, research assistant, pharmacist, study coordinator, other study site staff or relative of study site staff thus considered directly involved in the conduct of the study;
* Current addition/abuse of alcohol or drugs;
* Patients with any mental condition rendering them unable to understand the nature, scope, and possible consequences of the study;
* Pregnant or breast-feeding women;
* Patients living too far from investigational center or other conditions reducing the adherence to the protocol; Subjects unlikely or unable to comply with the Protocol requirements (e.g. illiterate, uncooperative, unable to return for follow-up visit, unable to use BGStar unlikely to complete the study)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2012-06-27 (Actual); Primary Completion 2015-07-30 (Actual); Study Completion 2015-07-30 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c levels from baseline | baseline to 12 months

SECONDARY OUTCOMES:
Percentage of participants with HbA1c ≤7.0% | at 12 months and 24 months
Variation in body weight from baseline | at 12 months and 24 months
Variation in waist circumference from baseline | at 12 months and 24 months
Variation in blood pressure from baseline | at 12 months and 24 months
Variation in lipid profile from baseline | at 12 months and 24 months
Quality of life: SF12 (Health Survey) questionnaire | at 12 months and 24 months
ADDQOL (Audit of Diabetes-Dependent Quality of Life) | at 12 months and 24 months
DTSQ (Diabetes Treatment Satisfaction Questionnaire) | at 12 months and 24 months
ABIM-14 (American Board of Internal Medicine satisfaction questionnaire) | at 12 months and 24 months
PDM (Patient involvement in the Decision Making process) questionnaire | at 12 months and 24 months
PHCO (Patient Health Care Orientation) questionnaire | at 12 months and 24 months
Participants satisfaction with SMBG meter assessed by Visual Analog Scale (VAS) | at 12 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Science & Operations, Study Director — Sanofi
Locations (20):
- Italy (20):
  - Investigational Site Number 016, Andria (BA)
  - Investigational Site Number 011, Avezzano
  - Investigational Site Number 006, Bergamo
  - Investigational Site Number 002, Brescia
  - Investigational Site Number 022, Catania
  - Investigational Site Number 001, Cusano Milanino
  - Investigational Site Number 013, Livorno
  - Investigational Site Number 015, Lucca
  - Investigational Site Number 004, Mariano Comense
  - Investigational Site Number 017, Messina
  - Investigational Site Number 008, Milan
  - Investigational Site Number 018, Napoli
  - Investigational Site Number 021, Potenza
  - Investigational Site Number 020, Ragusa
  - Investigational Site Number 014, Ravenna
  - Investigational Site Number 012, Rimini
  - Investigational Site Number 009, Roma
  - Investigational Site Number 019, Terlizzi (BA)
  - Investigational Site Number 007, Torino
  - Investigational Site Number 003, Udine